CLINICAL TRIAL: NCT05681546
Title: Risk Factors of Inferior Alveolar Nerve Block Failure: a Dental Student-centered Study
Status: Completed | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Gokhan Gurses, Assistant Professor, Selcuk University
Other Study IDs: Selcuk03
Record Dates: First submitted 2022-12-26; First posted 2023-01-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Anesthesia, Local
Keywords: anesteshia failure; mandibular nerve; dental student

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational Group: The investigators are going to observe the risk factors about inferior alveolar nerve block anesthesia.

SUMMARY:
Inferior alveolar nerve block anesthesia is one of the most commonly used regional block anesthesia in dentistry. The factors that determine the success of this type of anesthesia which is applied so frequently, are not reported in the literature. It is to reveal and evaluate patient and dentist-based factors, especially in anesthesia applied by trainee dentists who have just learned this anesthesia block.

DETAILED DESCRIPTION:
In this study, the investigators are going to observe 200 IANB anesthesia in our clinic. The investigators will evaluate the class, right/left handed, gender and experience on inferior alveolar nerve block of dental student. The criteria the investigators will evaluate for the patient are as follows; gender, body mass index, ramus height, left/right side, and maximum mouth opening amount. The criterion for the success of anesthesia are lost lip sensation within 10 minutes, no complication related to anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* having an indication of mandibular first or second molar extraction,
* being between 18 and 50 years old,
* not having any nerve or nerve-related disease,
* having a mouth opening 35 millimeters and above,
* not having an infected or inflamed tooth for extraction,
* being cooperative,
* non-allergic to articaine
* being right-handed (for dental-students)
* being intern (for dental-students)

Exclusion Criteria:

* anesthesia-related complications,
* more than twice the needed needle insertion
* wishing to quit the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: In this study, the investigators are going to observe 320 IANB anesthesia in our clinic, which is the Oral and Maxillofacial Surgery Department of Selçuk University.
Sampling Method: Probability Sample
Enrollment: 340 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-09-17 (Actual)

PRIMARY OUTCOMES:
Patrient-BMI index | after 5 minutes, patrients come to our clinic and sit on the dental unit.
  Ask the patrients their weight and height then note that as their bmi index.This note guides us amount of bichat and how it affects the failure of block anesthasia.
Patrient-Height of mandibular ramus | after 5 minutes, patrients come to our clinic and sit on the dental unit.
  measuring of mandibular ramus on panoromic radyography from mandibular angulus to condylar head.
Patrient-Gender | after 5 minutes, patrients come to our clinic and sit on the dental unit.
  attending patrients sex
Patrient-Maximum mouth opening | after 5 minutes, patrients come to our clinic and sit on the dental unit.
  before the anesthasia, make the patrients open their mouth maximum then measure it from lower incisors incisal edge to upper incisors incisal edge.
Gender | after 5 minutes, patrients come to our clinic and sit on the dental unit.
  attending dental studens sex
Student-Class | after 5 minutes, patrients come to our clinic and sit on the dental unit.
  attending dental students in which period for the explanation of their experiment level
Dental student-Mandibular nerve block experience | after 5 minutes, patrients come to our clinic and sit on the dental unit.
  attending dental students in which period for the explanation of their experiment level
which side for the mandibular block anesthasia | after 5 minutes, patrients come to our clinic and sit on the dental unit.
  Does the side of anesthesia according to the hand used affect its success?

CONTACTS AND LOCATIONS:
Overall Officials: Gökhan Gürses, Study Chair — Selcuk University, Faculty of Dentistry
Locations (1):
- Selcuk University, Dentistry Faculty, Selçuklu, Konya, Turkey (Türkiye)

REFERENCES:
- [Background] Thangavelu K, Kannan R, Kumar NS. Inferior alveolar nerve block: Alternative technique. Anesth Essays Res. 2012 Jan-Jun;6(1):53-7. doi: 10.4103/0259-1162.103375. PMID 25885503
- [Background] Kohler BR, Castellon L, Laissle G. Gow-Gates technique: a pilot study for extraction procedures with clinical evaluation and review. Anesth Prog. 2008 Spring;55(1):2-8. doi: 10.2344/0003-3006(2008)55[2:GTAPSF]2.0.CO;2. PMID 18327969